CLINICAL TRIAL: NCT01784328
Title: The Use of the Peristeen Bowel Irrigation System for People With Cauda Equina Syndrome
Brief Title: Peristeen Bowel Irrigation System in Cauda Equina
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manitoba (Other)
Collaborators: Manitoba Spinal Cord Injury Research Committee (Unknown); Canadian Paraplegic Association (Other)
Responsible Party: Principal Investigator, Dr. Karen Ethans, Director, Spinal Cord Injury Rehabilitation Program, University of Manitoba
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2013
Record Dates: First submitted 2013-01-30; First posted 2013-02-05 (Estimated); Last update posted 2016-07-06 (Estimated); Status verified 2016-07

CONDITIONS: Cauda Equina Syndrome
Keywords: Peristeen Bowel Irrigation System; Cauda Equina Syndrome; Lower Motor Neuron Neurogenic Bowel
MeSH Terms: conditions — Cauda Equina Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Use of a bowel irrigation system (Other): Open label. No placebo use in this study. All volunteers will trial the bowel irrigation system. Eligible volunteers will be those patients who have failed conventional supportive bowel care.
  Interventions: Device: Peristeen Bowel Irrigation System

INTERVENTIONS:
Device: Peristeen Bowel Irrigation System — A complete system for bowel Irrigation to manage bowel dysfunction

SUMMARY:
To compare the Peristeen Anal Irrigation System with conservative bowel management in a prospective study among spinal cord injured patients with lower motor neuron neurogenic bowel dysfunction.

DETAILED DESCRIPTION:
People with spinal cord injury (SCI) often have severe problems with management of bowel function, including incontinence, impaction, lengthy bowel routines and extremely slow transit times.The anal irrigation system is a recently available system to help patients with bowel dysfunction empty their bowels by using pulse water irrigation. The system consists of a rectal balloon catheter, manual pump and water container.

ELIGIBILITY:
Inclusion Criteria:

* Male or female >18 years or older
* Cauda equina spinal injury at least 12 months previously, with lower motor neuron bowel dysfunction and at least one of the following symptoms:
* Spending 30 minutes or more attempting to defecate each day or every second day
* Episodes of fecal incontinence once or more per month
* Abdominal discomfort before or during defecation

Exclusion Criteria:

* Coexisting major unresolved physical problems due to the injury
* Performance of transanal irrigation on a regular basis
* Evidence of bowel obstruction or active inflammatory bowel disease
* History of cerebral palsy, stroke, multiple sclerosis or diabetic polyneuropathy
* Previous colorectal or perineal surgery(excluding minor surgery such as hemorrhoidectomy)
* Pregnancy or lactation
* Immunosuppression
* Prior implant for sacral nerve stimulation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2013-03; Primary Completion 2016-04 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Change from baseline on Cleveland Clinic Constipation Scoring System after 10 weeks of treatment | At baseline Visit and again after 10 weeks of treatment
  A scoring system with a range of 0-30, with 30 representing the most severe symptoms. Will be used for volunteers whose primary complaint at baseline is constipation.
Change from baseline on the St. Mark's Fecal Incontinence Grading System after 10 weeks of treatment. | At baseline and again after 10 weeks of treatment
  A Grading system with a range of 0-24, with 24 representing the most severe symptoms. This will be used for volunteers whose primary complaint at baseline is fecal incontinence.

SECONDARY OUTCOMES:
Change from baseline in The Neurogenic Bowel Dysfunction Score after 10 weeks of treatment | At baseline and again after 10 weeks of treatment
  A symptom score ranging from 0-47, where each symptom of neurogenic bowel is weighted concerning it's impact on quality of life. A score of 47 represents severe symptoms.
Change from baseline in a modified American Society of Colon and Rectal Surgeons fecal incontinence score after 10 weeks of treatment. | At baseline and again after 10 weeks of treatment
  Symptom-related Quality of Life Score
Change from baseline measurement of Colonic Transit Time (CTT)after 10 weeks of treatment | At baseline and again after 10 weeks of treatment.
  The Metcalf method will be used.At the screening visit,eligible volunteers will be given a 7-day bowel diary and 3 SitzMark capsules with instructions on how to complete the diary and when to take the capsules. Abdominal X-rays will be obtained on Day 4 and 7. The patient will repeat the diary, SitzMark capsules and X-rays during the last week of study treatment.
Change from baseline on a numeric box scale to measure bowel function, influence on daily activities, and general satisfaction after 10 weeks of treatment. | At baseline and after 10 weeks of treatment.
  Numeric box scales with a range of 1-10
Measurement of Influence of Current Bowel Management on Quality of Life | After 10 weeks of treatment
  A numeric box scale with a range of 0-10, with 0 representing great reduction and 10 representing great improvement.

CONTACTS AND LOCATIONS:
Overall Officials: Karen Ethans, MD, Principal Investigator — University of Manitoba
Locations (1):
- WRHA Health Sciences Centre Rehabilitation Hospital, Winnipeg, Manitoba, Canada